CLINICAL TRIAL: NCT06072274
Title: Efficacy of Virtual Reality Educational Program on Empathy and Attitudes Toward Dementia in Caregivers
Brief Title: Efficacy of VR Educational Program on Empathy and Attitudes Toward Dementia in Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: N202308052
Record Dates: First submitted 2023-09-27; First posted 2023-10-10 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Dementia; Caregiver Burden
MeSH Terms: conditions — Dementia; Caregiver Burden

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality dementia simulation with guided reflection (Experimental): A single 3-hour virtual reality (VR) dementia simulation delivered in three consecutive segments, each followed by guided small-group reflection.
  Interventions: Behavioral: Virtual reality dementia simulation with guided reflection
- Traditional dementia education (lecture) (Active Comparator): Traditional dementia education (lecture) of equal duration.
  Interventions: Behavioral: Traditional dementia education (lecture)

INTERVENTIONS:
Behavioral: Virtual reality dementia simulation with guided reflection — A single 3-hour VR dementia simulation delivered in three consecutive segments, each followed by guided small-group reflection.
  Arms: Virtual reality dementia simulation with guided reflection
Behavioral: Traditional dementia education (lecture) — Instructor-led lecture of equal duration
  Arms: Traditional dementia education (lecture)

SUMMARY:
This randomized controlled trial evaluated a single-session virtual reality (VR) dementia simulation with guided small-group reflection compared with a time-matched, instructor-led lecture. A total of 227 caregivers of people with a formal diagnosis of dementia were enrolled and randomized. Empathy and attitudes toward dementia were assessed at baseline, immediately after the session, and 1 month after the session. Caregiver burden and psychological distress were assessed at baseline and 1 month after the session.

DETAILED DESCRIPTION:
This study used a parallel, two-arm randomized controlled design to evaluate a VR-based dementia simulation for caregiver education. A total of 227 caregivers of people with a formal diagnosis of dementia were enrolled and randomized to either (1) a single 3-hour VR dementia simulation delivered in three consecutive segments, each followed by guided small-group reflection (intervention), or (2) an instructor-led dementia education lecture of equal duration (control). Empathy and attitudes toward dementia were assessed at baseline, immediately post-session, and 1 month post-session. Caregiver burden and psychological distress were assessed at baseline and 1 month post-session.

ELIGIBILITY:
Inclusion Criteria:

1. Over 20 years;
2. Speak Chinese;
3. Currently providing care to a person with a formal diagnosis of dementia (paid formal caregivers or unpaid family caregivers).

Exclusion Criteria:

1. Those who are unable to use VR devices due to certain physical or mental situations;
2. Those who have fear/disgust for VR devices;
3. Those who feel dizzy after using VR devices;
4. For family caregivers: the care recipient is currently residing in a care facility.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2023-12-09 (Actual); Primary Completion 2024-03-16 (Actual); Study Completion 2024-03-16 (Actual)

PRIMARY OUTCOMES:
Change in empathy, measured by Jefferson Scale of Empathy | Immediate post-session
  Empathy is one of the major outcomes which we expect to be improved after the VR education program on dementia. The Jefferson Scale of Empathy (JSE): This scale is used to assess the empathy in caregivers. It is rated on a Likert seven-point scale, with 1 indicating strongly disagree and 7 indicating strongly agree. The scale consists of 20 items and is divided into three major dimensions: perspective taking, compassionate care, and standing in the patient's shoes. The total score ranges from 20 to 140, with higher scores indicating a more positive level of empathy.
Change in empathy, measured by Jefferson Scale of Empathy at 1 month | 1 month post-session
  Empathy is one of the major outcomes which we expect to be improved after the VR education program on dementia. The Jefferson Scale of Empathy (JSE): This scale is used to assess the empathy in caregivers. It is rated on a Likert seven-point scale, with 1 indicating strongly disagree and 7 indicating strongly agree. The scale consists of 20 items and is divided into three major dimensions: perspective taking, compassionate care, and standing in the patient's shoes. The total score ranges from 20 to 140, with higher scores indicating a more positive level of empathy.
Change in attitude, measured by Approach to Dementia Questionnaire | Immediate post-session
  Approach is one of the major outcomes which we expect to be improved after the VR education program on dementia. The Approach to Dementia Questionnaire (ADQ) is used to assess attitudes toward dementia care. The questionnaire consists of two dimensions: hope and person-centeredness, with a total of 19 items. It is rated on a Likert five-point scale, with 1 indicating strongly disagree and 5 indicating strongly agree. The total score ranges from 19 to 95, with higher scores indicating a more positive attitude of caregivers toward dementia care.
Change in attitude, measured by Approach to Dementia Questionnaire at 1 month | 1 month post-session
  Approach is one of the major outcomes which we expect to be improved after the VR education program on dementia. The Approach to Dementia Questionnaire (ADQ) is used to assess attitudes toward dementia care. The questionnaire consists of two dimensions: hope and person-centeredness, with a total of 19 items. It is rated on a Likert five-point scale, with 1 indicating strongly disagree and 5 indicating strongly agree. The total score ranges from 19 to 95, with higher scores indicating a more positive attitude of caregivers toward dementia care.

SECONDARY OUTCOMES:
Change in Caregivers' burden, measured by Zarit Burden Interview | Baseline and 1 month post-session
  We also expect that caregivers' burden would be reduced after the VR education program on dementia. Zarit Burden Inventory (ZBI): Developed by Zarit et al. in 1980, this inventory is used to measure negative emotions and perceived stress experienced by caregivers in the caregiving process. The ZBI consists of 22 items, and each item is rated on a scale of 0 to 4 based on the frequency of occurrence, ranging from "never" to "routinely." The total score ranges from 0 to 88, with higher scores indicating a greater caregiver burden. Scores between 0 and 20 indicate no or minimal burden, scores between 21 and 40 indicate mild to moderate burden, scores between 41 and 60 indicate moderate to severe burden, and scores between 61 and 88 indicate severe burden.
Caregivers' mental health status, measured by Brief Symptom Rating Scale-5 | Baseline and 1 month post-session
  We also expect that caregivers' mental health status would be improved after the VR education program on dementia. The BSRS-5 is a concise self-administered questionnaire adapted from the 50-item brief symptom rating scale. It assesses anxiety, depression, hostility, interpersonal sensitivity, and other symptoms, with scores for each item ranging from 0 to 4. A total BSRS-5 score exceeding 14 or a score of 1 or more on the suicide survey item may signal a severe mood disorder. Scores between 10 and 14 suggest moderate mood disorders, while scores between 6 and 9 may indicate mild mood disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Bai, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan